CLINICAL TRIAL: NCT06867731
Title: Endosonographic Shear Wave Elastography to Assess Liver Fibrosis
Brief Title: Endosonographic Shear Wave Elastography to Assess Liver and Splenic Fibrosis
Acronym: EUS SWE liver
Status: Enrolling by invitation | Type: Observational
Sponsor: Providence Medical Research Center (Other)
Collaborators: Fujifilm (Industry)
Responsible Party: Principal Investigator, Divyanshoo Kohli, Physician, Providence Medical Research Center
Other Study IDs: 2024000651
Record Dates: First submitted 2025-02-14; First posted 2025-03-10 (Actual); Last update posted 2025-05-30 (Actual); Status verified 2025-05

CONDITIONS: Liver Fibrosis; Cirrhosis
Keywords: Liver Fibrosis; Elastography; Liver Biopsy; Shear Wave Elastography; Endosonographic Shear Wave Elastography
MeSH Terms: conditions — Liver Cirrhosis; Fibrosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

GROUPS / COHORTS (1):
- Elastography: Diagnostic test: Endosonographic shear wave elastography
  Interventions: Procedure: Endosonographic Elastography; Diagnostic Test: Endosonographic shear wave elastography

INTERVENTIONS:
Procedure: Endosonographic Elastography — The patient will undergo a standard-of-care endoscopic ultrasound with liver biopsy. At the time, elastography of the liver and spleen will be performed while using the echoendoscope. Different degrees of pressure will be applied while performing elastography of the left and right lobes of the liver as well as the spleen. The E values and VsN values will be recorded and then compared to liver histology.
Diagnostic Test: Endosonographic shear wave elastography — The patient will undergo an upper endoscopic ultrasound procedure. During this procedure, the patient will be put to sleep and a trained endosonographer physician will insert an echo-endoscope through the mouth and guide it down to the stomach and the duodenum. This endoscope is equipped with technology that uses sound waves to assess the stiffness of the liver and spleen. For research purposes, the doctor will also press on these organs in order to take the additional measurements.

SUMMARY:
The study is being done to collect information on the effectiveness of endosonographic elastography (a technique which uses sound waves) to measure the stiffness of the liver and spleen. Investigators are trying to determine if shear wave elastography is a good way to measure fibrosis instead of biopsy.

DETAILED DESCRIPTION:
Study design This is a single-center, prospective, non-randomized, comparative study which will compare the diagnostic accuracy of Endoscopic ultrasound guided shear wave elastography (EUS-SWE) with liver biopsy for liver fibrosis.

Patients who will undergo a standard-of-care EUS guided liver biopsy (or have clinically obvious liver cirrhosis) will be prospectively enrolled after obtaining informed consent. All enrolled patients will undergo EUS guided liver biopsy, unless they have an obvious diagnosis of cirrhosis. EUS-SWE of the liver and spleen.

In selected patients who have been referred for EUS PPG measurement in addition to EUS liver biopsy, portal pressures will be measured as well and correlated with elastography of the spleen.

The patients will be initially assessed for need for liver biopsy by the gastroenterology/hepatology team as per the current standard of care. Only patients with a clear clinical indication for liver biopsy will be enrolled for the study.

Per current standard of practice at Providence Sacred Heart Medical Center, patients who need liver biopsy are referred to the interventional GI service for the procedure. These patients will be offered participation in the trial prior the endoscopic procedure. This detailed discussion will include participation in the study, background of the proposed study, inclusion and exclusion criteria, benefits and risks of the procedures and follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years (irrespective of sex)
* Patients determined clinically to have liver cirrhosis needing EUS for other reasons
* Patients determined clinically to be candidates for EUS guided liver biopsy
* Elevated liver enzymes without obvious etiology
* Clinical concern for cirrhosis requiring histological confirmation
* Patients with known cirrhosis without diagnostic dilemma
* Ability to provide informed consent and willing to participate

Exclusion Criteria:

* Surgically altered foregut anatomy which precludes safe endoscopic liver biopsy
* Coagulopathy with INR greater than 1.6 in patients on anticoagulant therapy
* Thrombocytopenia with platelet count less than 50,000/mL
* Pregnancy (positive urine pregnancy test in females of childbearing age)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing standard-of-care upper endoscopic ultrasound for liver biopsy or for other interventions in patients with known cirrhosis
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2025-01-30 (Actual); Primary Completion 2026-01-30 (Estimated); Study Completion 2027-01-30 (Estimated)

PRIMARY OUTCOMES:
Degree of fibrosis | Enrollment to 4 weeks
  Assessment of shear wave elastography as a surrogate for histological grade of liver fibrosis

SECONDARY OUTCOMES:
Comparative lobar pressure | Enrollment to 4 weeks
  Compare elastography values with standard or increased pressure
Spleen elasticity | Enrollment to 4 weeks
  Correlation of splenic elastography with portal pressures

CONTACTS AND LOCATIONS:
Overall Officials: Divyanshoo R Kohli, MD FACG FASGE, Principal Investigator — Providence Sacred Heart Medical Center
Locations (1):
- Providence Sacred Heart Medical Center, Spokane, Washington, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kohli DR, Mettman D, Andraws N, Haer E, Porter J, Ulusurac O, Ullery S, Desai M, Siddiqui MS, Sharma P. Comparative accuracy of endosonographic shear wave elastography and transcutaneous liver stiffness measurement: a pilot study. Gastrointest Endosc. 2023 Jan;97(1):35-41.e1. doi: 10.1016/j.gie.2022.08.035. Epub 2022 Aug 29. PMID 36049537